CLINICAL TRIAL: NCT07187518
Title: A Cross-sectional, Single-cohort, Bi-centre Clinical Investigation to Estimate Surrogate Bone Mineral Density (BMD) in Young and Middle-aged Men and Women Using Quantitative Ultrasound Imaging (POROUS)
Brief Title: Clinical Study to Estimate Bone Mineral Density With the POROUS Ultrasound Device
Acronym: POROUS-BMD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: POROUS GmbH (Industry)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R4C-BMD-01; 13GW0807 (Other Grant/Funding Number: BMBF)
Record Dates: First submitted 2025-09-15; First posted 2025-09-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Healthy; Osteopenia; Osteoporosis
Keywords: Osteoporosis; Osteopenia; Bone Tissue; Diagnostic Imaging; Ultrasound; Ultrasonography; Ultrasonic Diagnosis; DEXA Scan; DXA Scan; Dual X-Ray Absorptiometry; Bone Fractures; Osteoporotic Fractures; Hip Fractures; Spinal Fractures; Bone Mineral Density
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Fractures, Bone; Osteoporotic Fractures; Hip Fractures; Spinal Fractures | interventions — Weights and Measures

STUDY DESIGN:
Intervention Model Description: Comparative, single-cohort, interventional study model: investigational device vs. comparator device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BMD estimation in young and middle-aged men and women (Experimental): All participants are examined with the investigational device (POROUS R4C ultrasound device) and a comparator device (DXA).
  Interventions: Device: Measurements with the POROUS R4C ultrasound device at the midshaft tibia; Device: DXA measurement of the hip and lumbar spine

INTERVENTIONS:
Device: Measurements with the POROUS R4C ultrasound device at the midshaft tibia — The POROUS R4C ultrasound device measures the cortical bone of the midshaft tibia. Ultrasound gel is first applied onto the skin surface, covering the region of interest, followed by placing the ultrasound transducer with a medical ultrasound gel pad placed in front of it. At the marked position on the leg, four technical measurement readings are performed: 2x CortBS and 2x Multifocus, with repositioning the probe between individual measurements, the chronological order of which is not crucial. Scanning time for each measurement takes 1-2 minutes. Out of the four measurements, the two optimal measurements (one for CortBS and one for Multifocus) are selected by the device, based on pre-defined quality criteria.
Device: DXA measurement of the hip and lumbar spine — The following DXA measurements are to be performed: • Spine L1-4 • Hip left • Hip right (alternatively, if a valid measurement of the left hip is not possible) Scanning takes approximately 15 minutes. A maximum number of one repeat measurement is planned (e.g., hip or spine). Note: The DXA scan of the hip is performed on the same side of the body as the POROUS R4C ultrasound scan.

SUMMARY:
Osteoporosis is a widespread medical condition among older people. It causes the bones to weaken and become more likely to break. Osteoporosis and bone fracture risk are currently evaluated by looking at clinical risk factors and measuring bone mineral density (BMD). The lower the BMD is, the higher the risk of osteoporotic fractures in the future. An X-ray device called DXA is the main tool used to diagnose osteoporosis and fracture risk clinically. DXA measures two-dimensional BMD in the hip and spine. However, DXA devices are often not readily available at the point of care.

The POROUS ultrasound device offers a different approach by measuring various properties of the outer layer of the bone in the lower leg. It has several advantages over DXA: (1) higher and three-dimensional image resolution; (2) the ability to measure bone properties without radiation; (3) portability, it is a mobile medical device; 4) lower operational costs.

For this clinical study, we will recruit men and women between the ages of 21 and 55. Most of these study participants will not have evident clinical risks for osteoporosis. The goal for including this age group is to estimate the range of BMD values for younger people before BMD declines with age. In a separate clinical study, we are recruiting older participants. The study is anticipated to last one year.

Our major research questions are:

* Can the POROUS ultrasound device estimate BMD?
* How does its performance compare to DXA?
* What is the safety of the new device?

The participants will:

* answer questions about their medical history.
* be measured for height and weight.
* be examined with the two devices, DXA and POROUS.

DETAILED DESCRIPTION:
Medical background and current standard of care:

Osteoporosis is defined as a systemic skeletal disease characterized by low mineral bone mass and microarchitectural deterioration of bone tissue (Consensus Conference, 1994). This increased bone fragility is associated with susceptibility to fractures, which have substantial economic and societal burdens. Osteoporosis is routinely diagnosed through bone density assessments; however, there is a shortage of accurate means to characterize bone microstructure for diagnostic purposes. The POROUS R4C ultrasound device is capable of providing such information in detail.

The current standard of care (SoC) physical bone parameter for examining bone health is areal BMD (aBMD), typically measured by dual-energy X-ray absorptiometry (DXA) at the hip or spine. Scaling is given to score the patient's aBMD in comparison to a reference of a healthy bone. The resulting T Score compares the patient's aBMD to the peak aBMD of young adults of the same sex, while the Z score compares it to the average aBMD of the same age and sex. According to the operational WHO definition (1994), a T Score of -1.0 or above is considered normal, while scores between -1.0 and -2.5 indicate osteopenia, and scores of -2.5 or lower indicate osteoporosis.

The rationale for the clinical investigation:

Quantitative ultrasound (QUS) devices have several substantial advantages over X-ray-based technologies: a better safety profile (non-ionizing radiation), cost-efficiency, usability, and portability. These advantages can result in improved accessibility at point-of-care. The major challenge is, nonetheless, clinical performance. QUS devices that assess bone health have demonstrated varying performance in estimating surrogate aBMD values. aBMD estimation is calculated by empirical correlation with DXA reference measurements using a combination of ultrasound parameters and anthropometric information. We follow these clinical performance standards for aBMD estimation using the investigational POROUS R4C ultrasound device.

The investigational device:

The POROUS R4C is a non-invasive QUS device for measuring and quantifying microstructural, acoustic, and viscoelastic properties in cortical bone (e.g., in the tibia of the lower limb). The device can be used to acquire single-channel raw data in a pulse-echo mode and perform innovative signal processing and imaging techniques to determine physical bone biomarkers. Examples of physical bone biomarkers are cortical thickness and the speed of sound in the radial direction using refraction-corrected image reconstruction and frequency-dependent attenuation and pore-size distribution using spectral backscatter analysis. The measurement data are recorded by the acquisition software, and the post-processing analysis is done using separate algorithms. In pre-clinical and clinical studies (completed, ongoing, or planned), the effectiveness of spectral ultrasound backscatter analysis and refraction-corrected image reconstruction methods are being evaluated to assess bone quality, health, and biomechanical competence. In first-in-human pilot studies, the POROUS technology has demonstrated the feasibility of measuring cortical bone properties and estimating aBMD in smaller cohorts of participants.

The overall purpose of the clinical investigation:

In this confirmatory clinical investigation, data will be collected to characterize cortical bone properties and calculate surrogate aBMD values for young and middle-aged (21 to 55 years) men and women. In a separate confirmatory clinical investigation (POROUS-preFX, NCT06567054), data will be collected to characterize cortical properties and calculate surrogate aBMD values in older men and women (56 to 85 years). Together, the combined data will represent a broader range of estimated surrogate aBMD values and generate a POROUS T score for diagnostic purposes.

Clinical investigation design:

This is a cross-sectional, single-cohort, age- and sex-stratified study of participants aged 21 to 55 years. The rationale for selecting this age range is to gather data for this age group, while data from older participants are gathered in an independent clinical investigation (POROUS-preFX, NCT06567054).

Participants will be enrolled into different groups based on their age (consisting of five-year bands) and sex (males or females). All participants will undergo measurements using the investigational POROUS R4C ultrasound device and the comparator DXA device. Prior knowledge of aBMD values, whether measured by DXA or another type of bone densitometer, will not be recorded to avoid selection bias. The final analysis of study results will incorporate measured POROUS parameters (e.g., cortical thickness, cortical bone pore diameter distribution, cortical bone frequency-dependent ultrasound attenuation, cortical bone backscatter coefficient, speed of sound in the radial direction), anthropometric information (weight, height, BMI, sex), and age will be used to create a multivariate partial least squares (PLS) model to predict DXA-derived aBMD. This prediction model will be similar to the one described in the pilot studies (Armbrecht et al., JBMR Plus, 2021; Dehnen et al., Front Endocrinol, 2024). However, the formula will be re-developed based on the results of this study. The predictions will be made with DXA-derived aBMD values of the femur neck, total proximal femur, and lumbar spine collected in this study. Cross-calibration of DXA devices from different manufacturers will be done if necessary.

The participants will also receive a questionnaire regarding their medical history and any medications that may impact bone health.

Primary objective:

• To assess the performance of the POROUS R4C ultrasound device in estimating surrogate aBMD values (total femur).

Secondary objectives:

* To assess the performance of the POROUS R4C ultrasound device in estimating surrogate aBMD values (femoral neck and lumbar spine).
* To assess the safety of the POROUS R4C ultrasound device by monitoring adverse events affecting participants or healthcare professionals using the device.

Exploratory objectives:

* To generate T-score and Z-score scales (total femur, femoral neck, and lumbar spine) for the POROUS R4C ultrasound device and assess their performance.
* To collect data on cortical bone properties measured by POROUS R4C ultrasound device in young and middle-aged men and women.
* To assess the reproducibility of direct measurements by the POROUS R4C

Participants:

The clinical investigation will include 350 female and male participants. Prior knowledge of bone health or aBMD values will not be considered an enrolment criterion. All participants will undergo measurement using the investigational POROUS R4C ultrasound device at the midshaft tibia and a comparator DXA device at the total femur, femoral neck, and lumbar spine. The participants are stratified according to sex and age stratification into five-year bands:

* Age group 21-25, males/females = 25 per group, total = 50.
* Age group 26-30, males/females = 25 per group, total = 50.
* Age group 31-35, males/females = 25 per group, total = 50.
* Age group 36-40, males/females = 25 per group, total = 50.
* Age group 41-45, males/females = 25 per group, total = 50.
* Age group 46-50, males/females = 25 per group, total = 50.
* Age group 31-55, males/females = 25 per group, total = 50.

Screened and eligible individuals will be enrolled in the investigation until the necessary sample size for his/her corresponding group (based on age and sex) has been reached (see Table above). To avoid over-recruiting, once the necessary sample size for one group has been reached, no further individuals with matching age band or sex will be enrolled in the investigation.

Duration of the clinical investigation:

The planned overall clinical investigation is expected to last up to 12 months, from the first participant's enrolment until the last participant's clinical assessment. However, if the last participant's assessment is completed before the 12-month mark, the Sponsor may choose to conclude the investigation earlier.

Clinical procedures:

The following clinical procedures are performed during the investigation:

Screening:

* Inclusion/exclusion criteria
* Enrolment into corresponding age and sex groups.
* Informed consent

Clinical assessments:

* Measuring with the POROUS R4C ultrasound device at the central antero-medial tibia region
* Scanning with DXA (aBMD of the lumbar spine and proximal femur).
* Assessment of medical conditions and concomitant medication using a questionnaire.
* Recording of adverse events.

ELIGIBILITY:
Inclusion criteria:

* Female or male individuals aged 21 to and including 55 years.
* Written informed consent has been obtained.

Exclusion criteria:

* Presence of diseases that rule out valid measurements with the DXA and POROUS R4C ultrasound devices (e.g., fractures or metal implants in the examined bones, paralysis of the lower extremities, severe bone abnormalities).
* Open wounds or skin infections at the measurement site of the POROUS R4C ultrasound device.
* Inability to undergo the investigations required by the Clinical Investigation Plan (CIP) or cognitive limitations that preclude understanding of the Participant Information Sheet and the Informed Consent Document.
* Pregnancy and breastfeeding
* Individual is in custody by order of an authority or a court of law.
* Close affiliation with an investigational site, e.g., employment at an investigational site, close relative of an investigator, or dependent person (e.g., student of the investigational site).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-13 (Estimated)

PRIMARY OUTCOMES:
Primary Clinical Endpoint - POROUS | 12 months
  Assessment of the POROUS R4C ultrasound device in estimating surrogate aBMD values (total femur). The primary endpoint aims to obtain a statistically significant correlation between the surrogate POROUS-aBMD values and the respective DXA-aBMD values (total femur). Outcome measure: POROUS-aBMD (g/cm^2).
Primary Clinical Endpoint - DXA | 12 months
  Outcome measure: DXA-aBMD values - total femur (g/cm^2)

SECONDARY OUTCOMES:
Secondary Clinical Endpoint - POROUS | 12 months
  Assessment of the POROUS R4C ultrasound device in estimating surrogate aBMD values (femoral neck and lumbar spine). The secondary endpoint aims to obtain a statistically significant correlation between the surrogate POROUS-aBMD values and the respective DXA-aBMD values (femoral neck and lumbar spine). Outcome measure: POROUS-aBMD (g/cm^2).
Secondary Clinical Endpoint - DXA | 12 months
  Outcome measure: DXA-aBMD values - femoral neck and lumbar spine (g/cm^2)
Safety Endpoint: Incidence of procedural/device-related adverse events | 12 months
  In order to establish that the POROUS R4C ultrasound device is safe with a minimal number of adverse events affecting the participants or the healthcare professionals using the device, the following safety endpoints are investigated: • Incidence of procedural/device-related adverse events caused by the o Absorbed energy o Probe/transducer heating o Irritation by ultrasound gel o Release of substances o Inappropriate hygiene measures. • Other (serious) adverse events.

OTHER OUTCOMES:
Cortical bone properties: ultrasound cortical sound velocity in the radial direction | 12 months
  Outcome measure: ultrasound cortical sound velocity in the radial direction (m/s)
Cortical bone properties: cortical thickness | 12 months
  Outcome measure: ultrasound cortical thickness (mm)
Cortical bone properties: ultrasound frequency-dependent attenuation coefficient | 12 months
  Outcome measure: ultrasound frequency-dependent attenuation coefficient (dB)
Cortical bone properties: ultrasound frequency-dependent attenuation coefficient, intercept value of linear fit | 12 months
  Outcome measure: ultrasound frequency-dependent attenuation coefficient, intercept value of linear fit (dB/mm)
Cortical bone properties: ultrasound frequency-dependent attenuation coefficient, slope value of linear fit | 12 months
  Outcome measure: ultrasound frequency-dependent attenuation coefficient, slope value of linear fit (dB/MHz/mm)
Cortical bone properties: ultrasound cortical pore diameter distribution | 12 months
  Outcome measure: ultrasound cortical pore diameter distribution (μm)
Cortical bone properties: ultrasound backscatter coefficient | 12 months
  Outcome measure: ultrasound backscatter coefficient (dB)
Age | 12 months
  Outcome measure: age (years)
Sex | 12 months
  Outcome measure: sex (binary answer - m/f)
Weight | 12 months
  Outcome measure: weight (kg)
Height | 12 months
  Outcome measure: height (m)
BMI | 12 months
  Outcome measure: BMI (kg/m^2)
Performance Endpoint - POROUS T Score | 12 months
  Generation of T-score scales (total femur, femoral neck, and lumbar spine) for the POROUS R4C ultrasound device. The exploratory endpoint aims to obtain a statistically significant correlation between the surrogate POROUS-T scores and the respective DXA-T scores (total femur, femoral neck, and lumbar spine). Outcome measure: POROUS T Score (units on scale).
Performance Endpoint - DXA T Score | 12 months
  Outcome measure: DXA T Score - total femur, femoral neck, and lumbar spine (units on scale).
Performance Endpoint - POROUS Z Score | 12 months
  Generation of Z-score scales (total femur, femoral neck, and lumbar spine) for the POROUS R4C ultrasound device. The exploratory endpoint aims to obtain a statistically significant correlation between the surrogate POROUS-Z scores and the respective DXA-Z scores (total femur, femoral neck, and lumbar spine). Outcome measure: POROUS Z Score (units on scale).
Performance Endpoint - DXA Z Score | 12 months
  Outcome measure: DXA Z Score - total femur, femoral neck, and lumbar spine (units on scale).
Short-term intra-operator precision | 12 months
  The reproducibility of direct measurements by the POROUS R4C ultrasound device is assessed on 20 random participants: Two consecutive measurement acquisitions by the same operator (user) on the same participant. Outcome measure: coefficient of variation (%).
Short-term inter-operator repeatability | 12 months
  The reproducibility of direct measurements by the POROUS R4C ultrasound device is assessed on 20 random participants: Two measurement acquisitions by two operators (users) on the same participant on the same day. Outcome measure: coefficient of variation (%).
Long-term intra-operator precision | 12 months
  The reproducibility of direct measurements by the POROUS R4C ultrasound device is assessed on 20 random participants: Two measurement acquisitions by the same operator (user) on the same participant one month apart. Outcome measure: coefficient of variation (%).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Armbrecht, MD, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Department of Endocrinology and Metabolism, Charité Universitätsmedizin Berlin, Campus Mitte, Berlin
  - Centre of Muscle and Bone Research (ZMK), Charité Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dehnen C, Galindo A, Hoff P, Palme O, Maurer L, Raum K, Wiebe E. Quantitative ultrasound imaging reveals distinct fracture-associated differences in tibial intracortical pore morphology and viscoelastic properties in aged individuals with and without diabetes mellitus - an exploratory study. Front Endocrinol (Lausanne). 2024 Dec 16;15:1474546. doi: 10.3389/fendo.2024.1474546. eCollection 2024. PMID 39736865
- [Background] Armbrecht G, Nguyen Minh H, Massmann J, Raum K. Pore-Size Distribution and Frequency-Dependent Attenuation in Human Cortical Tibia Bone Discriminate Fragility Fractures in Postmenopausal Women With Low Bone Mineral Density. JBMR Plus. 2021 Sep 2;5(11):e10536. doi: 10.1002/jbm4.10536. eCollection 2021 Nov. PMID 34761144